CLINICAL TRIAL: NCT03061591
Title: Efficacy of Wholistic Turmeric Supplementation on Polyp Number and Size in Patients With Familial Adenomatous Polyposis A Randomized, Double Blinded, Placebo Controlled Study
Brief Title: Turmeric Supplementation on Polyp Number and Size in Patients With Familial Adenomatous Polyposis.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Head of Research and Development department, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-15-RK-0601-CTIL
Record Dates: First submitted 2017-02-14; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Familial Adenomatous Polyposis; FAP; FAP Gene Mutation
Keywords: Turmeric; Curcumin; colorectal polyps; colorectal neoplasia; mutyh mutation; apc mutation
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Intervention Model Description: 6 months of Curcumin vs. placebo treatment outcomes will be compared.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo and curcumin capsules are identical in appearance, and will be marked as "A" or "B". Study participants and staff will be blinded to the capsule content. A locked file containing the description will remain in a locked file on the study coordinators computer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wholistic Turmeric capsules (Active Comparator): Oral capsules of wholistic Turmeric capsules (Pukka herbs) (each capsule 100 mg curcumin) divided twice daily, or an identical placebo in 2 divided doses daily all taken before meals.
  Pukka's Wholistic Turmeric
  Interventions: Dietary Supplement: Wholistic Turmeric capsules
- Placebo (Placebo Comparator): Identical placebo capsules
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Wholistic Turmeric capsules — Oral capsules of wholistic Turmeric capsules (Pukka herbs) curcumin (each capsule 0.5100 m gr curcumin) for a total of 4 gr/d divided twice daily.
  Arms: Wholistic Turmeric capsules
Other: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
A Phase 2, randomized, double blind, placebo controlled trial for the effectivness of wholistic turmeric supplementation on polyp burden mong patients with Familial Adenomatouse Polyposis (FAP). Fourty Patients will be randomly assigned in a 1:1 ratio to recieve treatment with 8 capsuls (2*4 capsuls/day) of wholistic Turmeric capsules (Pukka herbs) or placebo for six months.

DETAILED DESCRIPTION:
Fourty individuals with identified APC mutation or MUTYH mutation that result in a phenotype of multiple colonic adenomas with or without duodenal adenomas will be included in the study. Participants will be allocated in a 1:1 ratio to receive either wholistic Turmeric capsules (Pukka herbs) or placebo for 6 months.

Participants will be assessed by a gastroenterologist 4-8 weeks after initiation, and at termination/conclusion visit at 6 months.

Blood, stool and urine samples will be collected at baseline, after 4-8 weeks and at 6 months just before final colonoscopy.

Serum samples will be used for testing complete blood count, liver function test, C-reactive protein (CRP) Various cytokines and small molecule measurements. Stool samples will be evaluated for microbiome composition.

Curcumin and curcuminoid levels will be measured in tissue serum, stool and urine will be measured in a subsample of patients.

Colonoscopy will be performed at study entry with removal of all polyps larger than 20mm, count and precise size measurement of polyps by a standard forceps, throughout the colon and in defined segments. Retained polyps will be counted and measured with an open forceps placed near the polyp to determine size. A full video and photos of the procedure will be taken. In cases with multiple polyps that cannot be counted or properly evaluated the PI will decide if a defined area like the rectum could be evaluated and will define it in terms of distance from the anus. In this case the video of the procedure will be evaluated by two separate gastroeneterologists blinded to treatment arm.

Frozen samples from normal mucosa will be taken at study entry. Samples from polyps will be taken preferably in cases with multiple polyp in order not to interrupt measurments.

Upper endoscopy only in patients with known duodenal adenomas will also be performed at study entry with as above evaluation. Sample from polyps and normal mucosa will be taken as above. A full video and photos of the upper endoscopy will be recorded as well.

A 2nd colonoscopy +/- gastroscopy will be performed at 6 months when all polyps will be counted and pictured by video and photography. Size determination in a similar way as above, throughout the colon or in the defined area as was decided at baseline colonoscopy.

Frozen samples from polyps and normal mucosa will be taken and polypoectomy will be performed upon the decision of the endoscopist in both lower and upper endoscopies.

Frozen tissue specimen will be used for H&E, various proliferation and apoptosis staining like KI67.

Tissue, blood, urine and stool samples will be frozen and sent for analysis.

Inclusion/screening visit will include:

1. Intake of patient medical history.
2. Exact documentation of identified genetic mutation per genetic consultation
3. Case report form (CRF).
4. Blood test including complete blood count, liver function test, C-reactive protein (CRP) and sera for subsequent cytokine analysis.
5. Urine and Stool collection .
6. Basline colonoscopy and/or upper endoscopy as detiled above with tissue collection and tattoo of tissue sampled.

Mid-term visit at 4-8 weeks will include:

1. Case report form (CRF).
2. Collection of Blood, urine and stool specimens.

Termination/conclusion visit will include:

1. Case report form (CRF).
2. Collection of blood, urine, stool specimens
3. Colonoscopy and upper endoscopy as described above with tissue collection of same tissue identified by tattoo.

ELIGIBILITY:
Inclusion Criteria:

1. An established clinical diagnosis of Familial Polyposis based on accepted clinical/ endoscopic and an identified APC or MUTYH mutation
2. Age 18-70 years.
3. Willing and able to give written consent.
4. At least 5 polyps, 2mm or lrager, with at least one larger then 4mm but not more then 20mm.
5. Colonic polyp burden that can be estimated by either counting or photographing(photo or video).

Exclusion criteria:

1. Pregnant or nursing women.
2. Stable does of any COX inhibitor drugs for more than 3 months prior to study entry,.
3. Concomitant severe or uncontrolled cardiovascular, hepatic, renal or metabolic disease.
4. Known allergy to curcumin.
5. Anticipated surgery within 6 months
6. Diagnosed polyps of high grade dysplasia or of adenocarcinomas in the GI on screening colonoscopy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Number of polyps | 6 months
Size of polyps | 6 months

SECONDARY OUTCOMES:
Histological apoptosis assays in frozen polyps and normal tissue (such as KI67, caspase 3 activity and COX-2 expression). | 6 months
Histological proliferation assays in frozen polyps and normal tissue (such as KI67, caspase 3 activity and COX-2 expression). | 6 months
Colonic microbiome composition, after curcumin therapy. | 6 months
Duodenal adenoma number. | 6 months
Duodenal adenoma size. | 6 months
Curcumin and curcuminoid levels in blood. | 6 months
Curcumin and curcuminoid levels in urine. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Revital Kariv, MD, Principal Investigator — Tel Aviv SMC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cruz-Correa M, Shoskes DA, Sanchez P, Zhao R, Hylind LM, Wexner SD, Giardiello FM. Combination treatment with curcumin and quercetin of adenomas in familial adenomatous polyposis. Clin Gastroenterol Hepatol. 2006 Aug;4(8):1035-8. doi: 10.1016/j.cgh.2006.03.020. Epub 2006 Jun 6. PMID 16757216
- [Background] Perkins S, Verschoyle RD, Hill K, Parveen I, Threadgill MD, Sharma RA, Williams ML, Steward WP, Gescher AJ. Chemopreventive efficacy and pharmacokinetics of curcumin in the min/+ mouse, a model of familial adenomatous polyposis. Cancer Epidemiol Biomarkers Prev. 2002 Jun;11(6):535-40. PMID 12050094
- [Background] Pettan-Brewer C, Morton J, Mangalindan R, Ladiges W. Curcumin suppresses intestinal polyps in APC Min mice fed a high fat diet. Pathobiol Aging Age Relat Dis. 2011;1. doi: 10.3402/pba.v1i0.7013. Epub 2011 Jun 1. PMID 22953026